CLINICAL TRIAL: NCT03636854
Title: Effect of Different Izotonic Quadriceps Exercise Training on Muscle Strength, Muscle Thickness and Balance in Healthy Individuals
Brief Title: Quadriceps Concentric vs Eccentric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Emrullah ALKAN, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ConEcc
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Muscle thickness; muscle strength; hop Test; Balance; performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentric Exercises (Experimental): 2 different concentric exercises will be done 3 times a week for 8 weeks.
  Interventions: Other: Concentric exercises
- Eccentric Exercises (Experimental): 2 different eccentric exercises will be done 3 times a week for 8 weeks.
  Interventions: Other: Eccentric exercises

INTERVENTIONS:
Other: Concentric exercises — Resistance concentric straight leg raise and knee extension will be done.
  Arms: Concentric Exercises
Other: Eccentric exercises — Resistance eccentric straight leg raise and knee extension will be done.
  Arms: Eccentric Exercises

SUMMARY:
The aim of the study is to compare the effects of concentric and eccentric exercises on muscle strength, muscle thickness and balance in healthy Individuals. Participants will randomly be divided into 2 groups: Concentric exercise (CE) group, eccentric exercise (EE) group. Concentric exercise group will be doing 2 concentric exercises and eccentric exercise group will be doing 2 eccentric exercise for 8 weeks. The evaluations will be repeated after 8 weeks of training to reveal the effects of concentric and eccentric exercises.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-25
* Healthy individuals
* Able to read, write and understand Turkish
* Willing and able to attend study

Exclusion Criteria:

* Any neurological, musculoskeletal or vascular disease in any of the lower extremity
* Having lower extremity musculoskeletal pain
* Previous history of surgery in any of the lower extremity
* Mental and cognitive disorders that would seriously affect cooperation

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Change in muscle thickness | Before training and after 8 weeks of training
  Change in muscle thickness will be measured by using Ultrasound

SECONDARY OUTCOMES:
Change in muscle strength | Before training and after 8 weeks of training
  Change in muscle strength will be assessed by using hand-held dynamometer.
Change in balance | Before training and after 8 weeks of training
  Change in balance will be measured by using Biodex Balance System.
Change in function | Before training and after 8 weeks of training
  Change in function will be measured by using single leg hop test

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No